CLINICAL TRIAL: NCT05380011
Title: Effects of Bimanual Task Training With and Without Constraint-Induced Movement Therapy on Upper Limb Functions in Hemiplegic Cerebral Palsy Children
Brief Title: Bimanual Task Training and Constraint-Induced Movement Therapy in Hemiplegic Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01263 Ayesha bint Ihsan
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Constraint Induced Movement Therapy; Bimanual Task Training; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: This will be single blinded study. The data will be coded and the analyst will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (CIMT and Bimanual Task Training) (Experimental): Constraint Induced Movement Therapy and Bimanual Task Training
  Interventions: Other: Constraint Induced Movement Therapy and Bimanual Task Training
- Group B (Bimanual Task Training) (Experimental): Bimanual Task Training
  Interventions: Other: Bimanual Task Training

INTERVENTIONS:
Other: Constraint Induced Movement Therapy and Bimanual Task Training — Constraint-Induced Movement Therapy and Bimanual Task Training will be performed. Constraint-Induced Movement Therapy has been shown to improve the uni-manual capacity of the impaired limb as well as improvement in quality and efficiency of movement and greater grasp function, whereas Bimanual Task Training has been shown to improve bimanual task performance, bilateral spontaneous use of affected limb and better bimanual coordination during daily life activities.
  Arms: Group A (CIMT and Bimanual Task Training)
Other: Bimanual Task Training — Bimanual Task Training will be performed. Bimanual Task Training has been shown to improve bimanual task performance, bilateral spontaneous use of affected limb and better bimanual coordination during daily life activities.
  Arms: Group B (Bimanual Task Training)

SUMMARY:
Various studies have been done comparing the individual effects of the two interventions of Constraint-Induced Movement Therapy and Bimanual Task Training in Hemiplegic Cerebral Palsy Children, but this study will compare the effects of combined interventions with a single intervention. This study will contribute to the upper motor function in hemiplegic cerebral palsy children i.e. manual dexterity, grasp and release function, quality and efficacy of movement, combined bimanual use of both hands and coordination, as a result of two intervention protocols.

DETAILED DESCRIPTION:
Various studies have been done comparing the individual effects of these two interventions of Constraint-Induced Movement Therapy and Bimanual Task Training in Hemiplegic Cerebral Palsy Children. But the literature comparing the effects of combined interventions of these two with either of the single intervention is sparse and limited, utilizing different clinical experiences and tools for the respective study. This study will contribute to the upper motor function in hemiplegic cerebral palsy children by comparing the effects of combined interventions with a single intervention with its overall effects in the respective population i.e. manual dexterity, grasp and release function, quality and efficacy of movement, combined bimanual use of both hands and coordination, as a result of two intervention protocols. A total of 54 patients diagnosed with Hemiplegic Cerebral Palsy will be selected for data collection according to the inclusion criteria. Patients will be divided into two groups, Group A and Group B. Group A will receive Bimanual Task Training and Constraint-Induced Movement Therapy (CIMT) and Group B will receive Bimanual Task Training alone. Constraint-Induced Movement Therapy (CIMT) will be performed 1.5 hours daily, with the constraint of 6 hours applied daily, thrice-weekly sessions, with a total of 10 to 12 sessions, for 4 weeks, along with, Bimanual Task Training with the practice of each task for 15 to 30 minutes, 1.5 hours daily, thrice-weekly sessions, with a total of 10 to 12 sessions, for 4 weeks respectively in Group A, whereas, Bimanual Task Training will be performed with the practice of each task for 15 to 30 minutes, 1.5 hours daily, thrice-weekly sessions, with a total of 10 to 12 sessions, for 4 weeks in Group B. Data will be collected at baseline, at 2 weeks and at 4 weeks after intervention from both groups. Upper Limb Functions will be measured using the Melbourne Assessment of Unilateral Upper Limb Function (MUUL) and Canadian Occupational Performance Measure (COPM) and Quality of life will be measured using Cerebral Palsy Quality Of Life measure (CP-QOL).

ELIGIBILITY:
Inclusion Criteria:

* Children with both Gender (Male and Female).
* Age between 5 to 15 years.
* Hemiplegic Cerebral Palsy Children.
* Patients fulfilling the criteria of Constraint Induced Movement Therapy (CIMT) i.e. wrist extension 20 degree, MCP and IP extension 10 degree.

Exclusion Criteria:

* Hemiplegic Cerebral Palsy children due to Traumatic Brain Injury.
* Patients having cognitive impairments.
* Hemiplegic Cerebral Palsy children with rigid deformities of upper extremity.
* Patients having associated Neurological Pathologies.
* Patients who are unable to follow treatment plan.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Melbourne Assessment of Unilateral Upper Limb Function (MUUL) | baseline
  Melbourne Assessment of Unilateral Upper Limb Function (MUUL) is considered one of the reliable tools to measure upper limb function. It consists of 16-items to measure the quality of unilateral upper limb function. Items of the assessment involve reach, grasp, and release. It shows excellent construct and inter-rater validity as well as its shows good reliability for treatment planning and clinical decision making. It has a total 16 number of items. Scoring is completed for 37 item sub-scores using a three, four or five-point scale and individually defined scoring criteria for each item. The maximum score is 122 and the minimum score is 0, where higher scores reflect the greater quality of upper limb movement.
Melbourne Assessment of Unilateral Upper Limb Function (MUUL) | 2 weeks
  Melbourne Assessment of Unilateral Upper Limb Function (MUUL) is considered one of the reliable tools to measure upper limb function. It consists of 16-items to measure the quality of unilateral upper limb function. Items of the assessment involve reach, grasp, and release. It shows excellent construct and inter-rater validity as well as its shows good reliability for treatment planning and clinical decision making. It has a total 16 number of items. Scoring is completed for 37 item sub-scores using a three, four or five-point scale and individually defined scoring criteria for each item. The maximum score is 122 and the minimum score is 0, where higher scores reflect the greater quality of upper limb movement.
Melbourne Assessment of Unilateral Upper Limb Function (MUUL) | 4 weeks
  Melbourne Assessment of Unilateral Upper Limb Function (MUUL) is considered one of the reliable tools to measure upper limb function. It consists of 16-items to measure the quality of unilateral upper limb function. Items of the assessment involve reach, grasp, and release. It shows excellent construct and inter-rater validity as well as its shows good reliability for treatment planning and clinical decision making. It has a total 16 number of items. Scoring is completed for 37 item sub-scores using a three, four or five-point scale and individually defined scoring criteria for each item. The maximum score is 122 and the minimum score is 0, where higher scores reflect the greater quality of upper limb movement.
Canadian Occupation Performance Measure (COPM) | baseline
  It is a client-centred outcome measure that helps the client to identify occupational performance issues and rates performance and satisfaction pre and post-intervention. This tool involves the first identification of problems or daily occupations of importance that are needed or expected to do, and then secondly, the client is asked to rate the importance of each occupation using a 10-point rating scale. In the third step. the client selects up to 5 most important problems to be addressed in intervention and the therapist enters the chosen problems and their importance ratings in the scoring section. In the fourth step, the client is asked to use a 10-point scale to rate their own level of performance and satisfaction with performance for 5 identified problems.
Canadian Occupation Performance Measure (COPM) | 2 weeks
  It is a client-centred outcome measure that helps the client to identify occupational performance issues and rates performance and satisfaction pre and post-intervention. This tool involves the first identification of problems or daily occupations of importance that are needed or expected to do, and then secondly, the client is asked to rate the importance of each occupation using a 10-point rating scale. In the third step. the client selects up to 5 most important problems to be addressed in intervention and the therapist enters the chosen problems and their importance ratings in the scoring section. In the fourth step, the client is asked to use a 10-point scale to rate their own level of performance and satisfaction with performance for 5 identified problems.
Canadian Occupation Performance Measure (COPM) | 4 weeks
  It is a client-centred outcome measure that helps the client to identify occupational performance issues and rates performance and satisfaction pre and post-intervention. This tool involves the first identification of problems or daily occupations of importance that are needed or expected to do, and then secondly, the client is asked to rate the importance of each occupation using a 10-point rating scale. In the third step. the client selects up to 5 most important problems to be addressed in intervention and the therapist enters the chosen problems and their importance ratings in the scoring section. In the fourth step, the client is asked to use a 10-point scale to rate their own level of performance and satisfaction with performance for 5 identified problems.
Cerebral Palsy Quality Of Life scale (CP-QOL) | baseline
  The Cerebral Palsy (CP) Quality Of Life scale-child is a condition-specific Quality Of Life (QOL) questionnaire designed for children with CP.
  Feasibility, sensitivity, Instrument validity and internal consistency of both self-and proxy-report questionnaires are good and are becoming a fundamental component of public health surveillance. QOL is broadly defined as a subjective multidimensional concept for assessing a person's wellbeing across numerous life indicators. The child self-report form contains 52 items and is divided into areas: well-being and social acceptance, functionality, participation and physical health, emotional well-being and self-esteem, access to services and pain and impact disability. All items are rated from 1 to 9, except for one item in the pain and impact disability domain, which is rated on a 5-point scale. All responses are then converted into scale scores between 0 to 100. Higher scores mean a higher quality of life and vice versa.
Cerebral Palsy Quality Of Life scale (CP-QOL) | 2 weeks
  The Cerebral Palsy (CP) Quality Of Life scale-child is a condition-specific Quality Of Life (QOL) questionnaire designed for children with CP.
  Feasibility, sensitivity, Instrument validity and internal consistency of both self-and proxy-report questionnaires are good and are becoming a fundamental component of public health surveillance. QOL is broadly defined as a subjective multidimensional concept for assessing a person's wellbeing across numerous life indicators. The child self-report form contains 52 items and is divided into areas: well-being and social acceptance, functionality, participation and physical health, emotional well-being and self-esteem, access to services and pain and impact disability. All items are rated from 1 to 9, except for one item in the pain and impact disability domain, which is rated on a 5-point scale. All responses are then converted into scale scores between 0 to 100. Higher scores mean a higher quality of life and vice versa.
Cerebral Palsy Quality Of Life scale (CP-QOL) | 4 weeks
  The Cerebral Palsy (CP) Quality Of Life scale-child is a condition-specific Quality Of Life (QOL) questionnaire designed for children with CP.
  Feasibility, sensitivity, Instrument validity and internal consistency of both self-and proxy-report questionnaires are good and are becoming a fundamental component of public health surveillance. QOL is broadly defined as a subjective multidimensional concept for assessing a person's wellbeing across numerous life indicators. The child self-report form contains 52 items and is divided into areas: well-being and social acceptance, functionality, participation and physical health, emotional well-being and self-esteem, access to services and pain and impact disability. All items are rated from 1 to 9, except for one item in the pain and impact disability domain, which is rated on a 5-point scale. All responses are then converted into scale scores between 0 to 100. Higher scores mean a higher quality of life and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- National Institute of rehabilitation medicine., Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No